CLINICAL TRIAL: NCT02736617
Title: A Phase II Study of Obinutuzumab (GA-101) in Combination With Ibrutinib (I) for the Treatment of Relapsed Mantle Cell Lymphoma
Brief Title: Obinutuzumab in Combination With Ibrutinib in Treating Patients With Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Stephen Spurgeon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015255; NCI-2016-00398 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00015255 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (obinutuzumab and ibrutinib) (Experimental): Patients receive obinutuzumab IV over 30 minutes on days 1, 8, and 15 of cycle 1, and day 1 of cycles 2-6. Patients also receive ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have PR continue to receive obinutuzumab IV every 2 months and ibrutinib PO QD for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Biological: Obinutuzumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759

SUMMARY:
This phase II trial studies how well obinutuzumab works in combination with ibrutinib in treating patients with mantle cell lymphoma that has returned (relapsed) or that does not respond to treatment (refractory). Obinutuzumab binds to a protein called cluster of differentiation (CD)20, which is found on B cells and some types of leukemia and lymphoma cells and help the immune system kill cancer cells. Ibrutinib blocks a protein called Bruton's tyrosine kinase (BTK), which may help keep cancer cells from growing. Giving obinutuzumab in combination with ibrutinib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Best overall response of complete response/partial response (CR/PR).

SECONDARY OBJECTIVES:

I. Toxicity defined as any adverse event (AE) grade 3 and higher. II. Progression free survival.

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. Gene expression profiling using Lymph5Cx test. II. Sequencing using the ion torrent platform (76 gene panel for known mutations in lymphoma).

III. Sequencing of BTK and phospholipase-C gamma (PLC) to evaluate for mutations.

IV. Minimal residual disease testing (MRD by flow cytometry and targeted sequencing post treatment).

OUTLINE:

Patients receive obinutuzumab intravenously (IV) over 30 minutes on days 1, 8, and 15 of cycle 1, and day 1 of cycles 2-6. Patients also receive ibrutinib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving partial response (PR) continue to receive obinutuzumab IV every 2 months and ibrutinib PO QD for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of relapsed or refractory mantle cell lymphoma as follows:

  * Diagnosis of mantle cell lymphoma (MCL) must include morphology and expression of either cyclin D1 in association with other relevant markers (eg, CD19, CD20, CD5) or evidence of t(11;14) as assessed by cytogenetics, fluorescent in situ hybridization (FISH), or polymerase chain reaction (PCR)
  * Relapsed or refractory disease is defined as no response or progressive disease to prior treatment if the prior treatment comprised any of the following:

    * 1 regimen containing an anti-CD20 antibody administered for >= 2 doses, and/or
    * >= 1 regimen containing 1 cytotoxic agent (e.g., bendamustine, chlorambucil, cyclophosphamide, cytarabine, doxorubicin) administered for 2 cycles
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma (Cheson Criteria); the site of disease must be greater than 1.5 cm in the long axis regardless of short axis measurement or greater than 1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1.0 K/cu mm; for subjects with ANC < 1.0 K/cu mm due to significant marrow involvement by MCL, ANC must be > .5 K/cu mm
* Platelets (plt) >= 50 K/cu mm; for subjects with plt < 50 K/cu mm due to significant marrow involvement by MCL, plt must be > 25 K/cu mm
* Total bilirubin =< 2.5 X institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine =< 2
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials; men must agree to not donate sperm during and after the study; for females, these restrictions apply for 18 months after last dose of obinutuzumab, or 1 month after the last dose of ibrutinib, whichever is later; for males, these restrictions apply for 180 days after the last dose of obinutuzumab or 3 months after the last dose of ibrutinib, whichever is later
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening; women who are pregnant or breastfeeding are ineligible for this study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Major surgery within 4 weeks of drug administration
* Diagnosed or treated for malignancy other than MCL, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 2 years
  * Adequately treated non-melanoma skin cancer or melanoma in situ without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Asymptomatic prostate cancer managed with "active surveillance"
  * Localized prostate cancer treated with definitive treatment including radiation or surgery. Patients on adjuvant hormone deprivation treatment such as lupron are eligible. Patients with known metastatic disease are ineligible
* History of stroke or intracranial hemorrhage within 6 months prior to randomization
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon)
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization
* Requires treatment with strong cytochrome P450 3A (CYP3A) inhibitors
* Subjects who have had standard cytotoxic chemotherapy or radiotherapy within 3 weeks prior to entering the study or those whose adverse events due to agents administered more than 3 weeks earlier have not recovered to =< grade 1; this excludes alopecia and hematologic adverse events
* Subjects who have had radiotherapy within 2 weeks prior to entering the study or those whose adverse events due to radiotherapy more than 2 weeks earlier have not recovered to =< grade 1
* Subjects who have received investigational or approved oral or "targeted" agents (such as spleen tyrosine kinase [SYK], phosphatidylinositol 3 kinase [PI3K], B-cell chronic lymphocytic leukemia [CLL]/lymphoma 2 [bcl-2], BTK inhibitors) or lenalidomide within 1 week prior to entering the study or those whose adverse events due to agents administered more than 1 week earlier have not recovered to =< grade 1; this excludes hematologic adverse events; the exception is subjects who are currently receiving ibrutinib (for < 14 days). In this case, ibrutinib can be continued
* Subjects who have received monoclonal antibodies (such as Rituxan) within 1 week prior to entering the study or those whose adverse events due to agents administered more than 1 week earlier have not recovered to =< grade 1; this excludes hematologic adverse events
* Subjects who are actively receiving any other investigational agents
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition as obinutuzumab or ibrutinib or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women are excluded from this study
* Known history of human immunodeficiency virus (HIV) or active hepatitis C
* Virus or active hepatitis B virus infection; patients who are hepatitis B core antibody (HBcAb) positive may be eligible as long as there is no evidence of active infection with negative hepatitis B (Hep B) by polymerase chain reaction (PCR); in this case, Hep B PCR must be monitored monthly
* Any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk
* Patients previously treated with ibrutinib > 14 days are ineligible; no drug intervention or cessation is required for patients already receiving ibrutinib prior to initiation of on-study therapy
* Active graft versus (vs.) host disease (GVHD)
* Ongoing glucocorticoids (prednisone > 10 mg daily, or equivalent); higher doses (> 10 mg daily) are permitted for up to 5 days to help control disease related symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Participants receive 1000mg Obinutuzumab intravenously (IV) over 30 minutes on days 1, 8, and 15 of cycle 1, and day 1 of cycles 2-6. Patients also receive ibrutinib once daily by mouth on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have at least partial response (PR) will continue to receive obinutuzumab IV every 2 months and oral ibrutinib for 2 years in the absence of disease progression or unacceptable toxicity.
Period: Treatment
Arm/Group | Overall Study
Started | 10
Completed | 7
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Period: Maintenance
Arm/Group | Overall Study
Started | 7
Completed | 2
Not Completed | 5
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants who receive at least one dose of either study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 72.0 [55.0 to 81.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 10
Disease status at enrollment [Count of Participants; unit: Participants] — Disease response to previous therapy was measured using the Lugano criteria as measured by fluorodeoxyglucose-positron emission tomography (FDG-PET). Stable disease means no metabolic response, with no significant change in FDG uptake from the previous therapy's baseline measure. Progressive disease means there was an increased intensity of FDG uptake over the previous baseline or the appearance of a new FDG-avid lesion.
  Participants
    Stable Disease | 5
    Progressive Disease | 5
Mantle Cell Lymphoma International Prognositic Index (MIPI) Risk Class [Count of Participants; unit: Participants] — Risk score for survival in patients with mantle cell lymphoma is a combination of age, Eastern Cooperative Oncology Group (ECOG) performance status at diagnosis, serum lactate dehydrogenase (LDH), white blood cell (WBC) count, and optional Ki-67 (proliferation marker) positivity percent. Risk is a 3-level score of High (bad), Intermediate, and Low (good).
  Participants
    Intermediate Risk | 3
    High Risk | 7
Ki-67 positivity, % (proliferation marker) [Median (Full Range); unit: percent positive nuclei in field] | 65 [10 to 90]
Eastern Cooperative Oncology Group (ECOG) at screening [Count of Participants; unit: Participants] — Six point scale measuring the ability of patients to tolerate therapies during serious illness based on symptoms and mobility. Ranges from a minimum of 0 (asymptomatic, best score) to a maximum of 5 (death)
  Participants
    ECOG 0 | 1
    ECOG 1 | 9
Months between diagnosis and enrollment [Median (Full Range); unit: Months] | 21.5 [3.4 to 116.9]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Best Overall Objective Response or Complete Response/Partial Response (CR/PR)
Description: Overall response is measured combining bone marrow biopsy with CT or PET, measuring target and evaluable non-targeted lesions, according to the Lugano criteria. For FDG-PET, the Deauville criteria is used in conjecture with CT to assess lesion FDG-update. Deauville scale ranges from 1 to 5, where 1 is best (no uptake or no residual uptake) and 5 is worst (markedly increased uptake or any new lesion). If bone marrow is involved prior to treatment, infiltrate must have cleared on repeat biopsy for CR; bone marrow assessment is irrelevant for determination of PR. Measurements are taken at baseline, end of cycle 2, end of induction (after cycle 6) and every 4 months thereafter. Best overall response is any CR or PR reported since start of therapy. Percent of participants with complete response or partial response (CR+PR) are reported along with 95% confidence interval.
Time Frame: From first dose of study therapy until the 6-month disease assessment (Cycle 6, Day1 or End of Induction Day 28). Disease assessment is also assessed at end of Cycle 2 (2-months).
Population: Efficacy evaluable population: those who receive at least one dose of both study drugs and had one response assessment (after cycle 2). Any patient who clinically progresses prior to their first scheduled response assessment will be included in the efficacy set and will be counted as a non-responder.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Efficacy Evaluable: Participants who receive at least one dose of both study drugs and have one response assessment (after cycle 2) are eligible for the efficacy evaluable set. Participants progressing prior to the first scheduled response assessment are counted as non-responders. Evaluable participants who do not have response assessments (e.g. are removed for toxicity) are also counted as non-responders. All other progressions must be confirmed by imaging. One participant withdrew consent 6 days after starting study therapy and was considered ineligible for the efficacy evaluable set.
Arm/Group | Efficacy Evaluable
Number analyzed (Participants) | 9
percentage of participants | 89 [62 to 100]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Median progression free survival is measured from first day of study therapy until disease progression or death, whichever comes first. Participants who progress prior to their first scheduled disease assessment are considered to have clinically progressed. Participants who do not progress are censored at the time of their last disease assessment. The Kaplan-Meier method is used to estimate median PFS. 95% confidence interval is provided, although upper limit was not achieved (insufficient number of progressions)
Time Frame: Time from the first day of combined study treatment to disease progression or death, whichever occurs first, assessed up to approximately 4 years, 11 months, after first dose of study drug(s)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efficacy Evaluable
Number analyzed (Participants) | 9
months | 14 [6.9 to NA] — Too few participants progressed to calculate the upper limit of the 95% confidence interval

3. Secondary Outcome: Number of Participants With Treatment-related Toxicities, Grade 3 or Higher, as Assessed by CTCAE v4.0
Description: Defined as any adverse event grade 3 or higher, classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0, from the first dose of study drug(s) until 30 days after the last dose of study drug(s)
Time Frame: Measured from the first dose of either study drug until 30 days after the last dose of study drug, for approximately 4 years, 11 months.
Population: All participants receiving at least 1 dose of IV Obinutuzumab or oral Ibrutinib
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 10
participants
  Infections and infestations | 1
  Infusion related reaction | 1
  Neutrophil count decreased | 4
  Platelet count decreased | 2
  Stroke | 1

ADVERSE EVENTS:
Time Frame: From the first dose of either IV Obinutuzumab or oral Ibrutinib until 30 days after the last dose, up to approximately 5 years (4 years, 11 months)
Description: All AE and SAE were collected and reporting, irrespective of grade or attribution. Given only 10 participants were enrolled we were unable to apply the 5% threshold on adverse events.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=10)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=10)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 4 (5)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 3 (7)
Fever (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (7)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (15)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Palpitations (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 4 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (7)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was powered to detect an 85% response rate compared to a 55% control rate. Simon's Two-Stage design planned to enroll 6 at Stage 1; if 4 or more achieved CR/PR then an additional 14 would be enrolled in Stage 2 for a total of 20 participants. Study satisfied Stage 1 requirements but lagging enrollment caused study to close with only 10 participants enrolled. Of the 10 only 9 were efficacy evaluable. Power: P(x>=8|n=9, p=0.85) = 0.599; x=success, n=evaluable, p=expected probability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT02736617/Prot_SAP_000.pdf